CLINICAL TRIAL: NCT03600142
Title: A Stigma Reduction Intervention at Time of Entry Into Antenatal Care to Improve PMTCT Services in Tanzania (Maisha)
Brief Title: A Stigma Reduction Intervention at Time of Entry Into Antenatal Care to Improve PMTCT Services in Tanzania
Acronym: Maisha
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Melissa Watt, Associate Professor of Population Health Sciences, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21TW011053-01 (NIH); 1R21TW011053-01 (NIH)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
Keywords: Stigma; HIV; Counseling; Tanzania; Pregnancy; Cognitive-behavioral therapy; Retention in care; Prevention of mother to child transmission
MeSH Terms: conditions — HIV Infections; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (No Intervention): Participants randomized to the control condition will receive the standard HIV counseling protocol in the clinic, which is administered by clinic nurses. According to the Tanzania PMTCT guidelines, HIV pre-test counseling should provide education about HIV and prepare a woman (and her partner, if present) for HIV testing. For anyone who tests positive for HIV, counseling should help the woman/couple to accept an HIV test result and discuss implications for treatment.
- SoC + stigma counseling (Maisha) (Experimental): Participants randomized to the intervention condition will receive the SoC counseling plus Maisha, a brief, scalable, theory-based counseling intervention that addresses HIV stigma at entry into antenatal care. Maisha involves a video delivered to all women prior to HIV testing, and, if a woman tests positive for HIV, two counseling sessions. If a male partner is present with the women, he may also be enrolled and participate in the first two counseling sessions together with the woman.
  Interventions: Behavioral: Mashia

INTERVENTIONS:
Behavioral: Mashia — Maisha is a brief, scalable, theory-based counseling intervention that addresses HIV stigma at entry into antenatal care. The intervention will be developed in a formative phase and includes 1) a video and counseling session prior to HIV testing that addresses HIV stigma, and 2) two post-test HIV counseling sessions for HIV-infected individuals, building on the video content to provide emotional support, address stigma, and reinforce the value of care engagement.
  Arms: SoC + stigma counseling (Maisha)

SUMMARY:
This study will pilot test a brief, scalable intervention called Maisha (Swahili for life), to address HIV stigma for women presenting to antenatal care in Tanzania and male partners who accompany them. The intervention will include: 1) a video and brief counseling that addresses HIV stigma at the start of the ANC visit (prior to HIV testing), and 2) two stigma-based counseling sessions for individuals who are HIV infected, building on the video content to provide emotional support, promote acceptance, address stigma, and reinforce care engagement. The primary intervention outcome is engagement in PMTCT care among women who are HIV infected. The investigators will also examine HIV stigma outcomes (enacted, anticipated, internalized) among all groups of participants, including individuals who are already established on ART and indiviudals who are HIV uninfected.

DETAILED DESCRIPTION:
HIV-related stigma has been identified as a significant reason for loss to follow up in prevention of mother-to-child transmission of HIV (PMTCT) programs. Antenatal care (ANC) provides a unique and important entry point to address HIV stigma. Stigma-based counseling during the first ANC visit can promote readiness to initiate or sustain treatment among those who are HIV infected, and can address stigmatizing attitudes and behaviors among those who are uninfected. We are proposing to pilot test a brief, scalable intervention called Maisha (Swahili for life), to address HIV stigma for women and their partners presenting to ANC in Tanzania. The intervention will include: 1) a video and brief counseling for women and their partners (if present) that addresses HIV stigma at the start of the ANC visit (prior to HIV testing), and 2) two stigma-based counseling sessions for women who are HIV infected, building on the video content to provide emotional support, promote acceptance, address stigma, and reinforce care engagement, with the opportunity for male partners to attend the first follow-up counseling session after testing. The primary intervention outcome is engagement in PMTCT care among women who are HIV infected. As a secondary outcome we will also look at linkage to HIV care among men who are HIV infected. We will also examine HIV stigma outcomes (enacted, anticipated, internalized) among all groups of people, including those who are already established on ART and those who are HIV uninfected. The intervention content is based on principles of cognitive-behavioral therapy (addressing automatic negative thoughts about the self, future and the world) to address and mitigate multiple forms of HIV stigma (internalized, anticipated and enacted). We will conduct a pilot RCT of the intervention, enrolling all women who attend a first ANC appointment at two clinics in the Moshi district. If women come to the ANC visit with a male partner, the partner will be invited to enroll as well. Maisha will be compared to the standard of care HIV counseling. In addition to a baseline assessment, all participants who are identified as HIV-infected and their partners will get a follow-up assessment three months after enrollment. A subset of participants who are identified as HIV-uninfected but who report high levels of HIV stigmatizing attitudes at baseline will also receive a follow-up assessment three months after enrollment. Measures will include health outcomes (care engagement, adherence, depression), stigma outcomes, and HIV disclosure. Quality assurance data will be collected and the feasibility and acceptability of the intervention and RCT will be described. Statistical analysis will examine differences between conditions in health outcomes and stigma measures, stratified by HIV status. We hypothesize that 1) among HIV infected individuals, individuals receiving the Maisha intervention will report better engagement in PMTCT care/linkage to HIV care and lower levels of internalized HIV stigma, as compared to individuals receiving the standard of care, and 2) among HIV uninfected individuals, individuals receiving the pre-test video and counseling will report lower levels of stigmatizing attitudes when compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* If female: Pregnant and attending first antenatal care (ANC) appointment for the current pregnancy at one of the two study sites
* If male: Accompanying an enrolled woman to her first ANC appointment.

Exclusion Criteria:

* Impaired mental status
* Does not speak Swahili

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1539 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Watt, PhD, Principal Investigator — University of Utah; Blandina Mmbaga, MD, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The data from the formative and pilot trial work in this R21 will be shared within the constraints required for the protection of confidentiality for study subjects. With a data transfer agreement from our Institutional Review Board, the investigators are willing to share raw data with researchers and program leaders from other institutions.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared starting 6 months after publication.
Access Criteria: Data will be shared with investigators who are interested in secondary data analysis or inclusion in meta-analyses. The investigators will work with individuals requesting data access to put in place an appropriate data transfer agreement. The study PI will review all requests for data sharing.

REFERENCES:
- [Background] Watt MH, Knettel BA, Knippler ET, Kisigo G, Ngocho JS, Renju J, Rogathi J, Sao SS, Minja L, Osaki H, Mwamba RN, Mmbaga BT. The development of Maisha, a video-assisted counseling intervention to address HIV stigma at entry into antenatal care in Tanzania. Eval Program Plann. 2020 Dec;83:101859. doi: 10.1016/j.evalprogplan.2020.101859. Epub 2020 Aug 5. PMID 32795711
- [Result] Watt MH, Minja L, Knettel BA, Mwamba RN, Osaki H, Ngocho JS, Kisigo GA, Renju J, Vissoci JRN, Sao SS, Mmbaga BT. Pilot Outcomes of Maisha: An HIV Stigma Reduction Intervention Developed for Antenatal Care in Tanzania. AIDS Behav. 2021 Apr;25(4):1171-1184. doi: 10.1007/s10461-020-03093-9. Epub 2020 Nov 12. PMID 33180253
- [Derived] Cohen SR, Marchand V, Calkins K, Stephens MJ, Barabara ML, Minja LM, Olomi GA, Mlay J, Mlay PS, Hanson OR, Mmbaga BT, Watt MH. Participatory simulation training design: The MAMA interprofessional team-training program for obstetric care of pregnant individuals living with HIV in Tanzania. Eval Program Plann. 2025 Jun;110:102550. doi: 10.1016/j.evalprogplan.2025.102550. Epub 2025 Jan 31. PMID 39914273
- [Derived] Watt MH, Knippler ET, Minja L, Kisigo G, Knettel BA, Ngocho JS, Renju J, Osaki H, Mwamba R, Rogathi JJ, Mmbaga BT. A counseling intervention to address HIV stigma at entry into antenatal care in Tanzania (Maisha): study protocol for a pilot randomized controlled trial. Trials. 2019 Dec 30;20(1):807. doi: 10.1186/s13063-019-3933-z. PMID 31888700

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SoC): Participants randomized to the control condition (n=773) received the standard HIV counseling protocol in the clinic, which was administered by clinic nurses. According to the Tanzania PMTCT guidelines, HIV pre-test counseling should provide education about HIV and prepare a woman (and her partner, if present) for HIV testing. For anyone who tested positive for HIV, counseling helped the woman/couple to accept an HIV test result and discuss implications for treatment.
- SoC + Stigma Counseling (Maisha): Participants randomized to the intervention condition (n=758) received the SoC counseling plus Maisha, a brief, scalable, theory-based counseling intervention that addresses HIV stigma at entry into antenatal care. Maisha involves a video delivered to all women prior to HIV testing, and, if a woman tested positive for HIV, two counseling sessions. If a male partner was present with the women, he was also enrolled and participated in the first two counseling sessions together with the woman.
  Mashia: Maisha is a brief, scalable, theory-based counseling intervention that addresses HIV stigma at entry into antenatal care. The intervention was developed in a formative phase and includes 1) a video and counseling session prior to HIV testing that addresses HIV stigma, and 2) two post-test HIV counseling sessions for HIV-infected individuals, building on the video content to provide emotional support, address stigma, and reinforce the value of care engagement.
Period: Overall Study
Arm/Group | Standard of Care (SoC) | SoC + Stigma Counseling (Maisha)
Started | 777 | 762
Completed | 773 | 758
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | SoC + Stigma Counseling (Maisha) | Total
Number analyzed (Participants) | 773 | 758 | 1531
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 26 [23 to 31] | 26 [22 to 30] | 26 [23 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 519 | 520 | 1039
  Male | 254 | 238 | 492
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 773 | 758 | 1531
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 773 | 758 | 1531
Had Secondary Education [Count of Participants; unit: Participants] | 319 | 316 | 635
Married [Count of Participants; unit: Participants] | 484 | 458 | 942
Employed [Count of Participants; unit: Participants] | 141 | 161 | 302
HIV Positive [Count of Participants; unit: Participants] | 31 | 35 | 66
Stigmatizing Attitudes [Count of Participants; unit: Participants] | 10 | 12 | 22
Anticipated Stigma [Count of Participants; unit: Participants] | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: HIV Care Engagement (Female HIV-infected Participants Only)
Description: For HIV-infected female participants, retention in care will be assessed via medical record review, with retention defined as having no more than a 60 day gap between PMTCT visits at the study clinic, or having record of an official transfer to another clinic.
Time Frame: Post-assessment (3 months after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | SoC + Stigma Counseling (Maisha)
Number analyzed (Participants) | 26 | 28
Participants | 3 | 3
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs SoC + Stigma Counseling (Maisha); We were aware that our resources of time and funding would not be sufficient to detect a significant difference in the HIV care outcome, and that we would only be able to detect observational signals of impact. We aimed for a minimum of 50 WLHIV, which is considered an adequate sample to assess feasibility and acceptability in a pilot intervention study. Given an estimated 5% HIV prevalence among women presenting for ANC, this required us to enroll 1000 female participants; Test type: Non-Inferiority — For WLHIV (n=55), chi-square tests were used to assess differences between conditions in the proportion of participants who were retained in HIV care at 3 months post enrollment; p = 0.963, Chi-squared

2. Primary Outcome: Attitudes Toward People Living With HIV, Blame/Judgement Subscale (HIV-uninfected Participants Only)
Description: Self-report, measured by a modified version of personal and attributed stigma scales (Visser, Kershaw, Makin, & Forsyth, 2008)
  Scoring: 6 items. Item scores range from 0-3 (Strongly Disagree to Strongly Agree). Item responses are totaled for a summary score. Total scores range 0-18, with higher scores indicating greater stigma.
Time Frame: Post-assessment (3 months after enrollment)
Population: A sub-set up individuals who were HIV-negative at baseline were invited to return for 3-month follow-up. Individuals with total stigmatizing attitude scores >14 were eligible for follow-up; of those who met criteria, a random 60% were invited for follow-up in order to reach a minimum sample powered to detect differences in HIV stigma.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | SoC + Stigma Counseling (Maisha)
Number analyzed (Participants) | 134 | 159
units on a scale | 6.4 (4.6) | 4.6 (4.0)

3. Other Pre Specified Outcome: Quality Assurance (QA Data)
Description: Quality assurance data will be collected on feasibility, acceptability, and fidelity of Maisha session to the intervention manual. Sessions will be recorded and a subset of recordings will be reviewed to assess whether core components of the sessions were completed. Follow-up surveys will include items on participant satisfaction with the intervention format, session content, and interventionist. A subset of participants will also be selected to give additional qualitative feedback.
Time Frame: Post-assessment (3 months after enrollment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months.
Description: The definition of adverse events and/or serious adverse events does not differ from the ClinicalTrials.gov definition.
Arm/Group | Standard of Care (SoC) | SoC + Stigma Counseling (Maisha)
All-Cause Mortality (participants affected / at risk) | 0/777 | 0/762
Serious Adverse Events (participants affected / at risk) | 0/777 | 0/762
Other Adverse Events (participants affected / at risk) | 0/777 | 0/762

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT03600142/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT03600142/ICF_002.pdf